CLINICAL TRIAL: NCT00783549
Title: A Study in Healthy Volunteers of Single Doses of Orally Administered GSK1292263 to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Compound Alone and When Co-administered With Sitagliptin
Brief Title: A Study in Healthy Volunteers of Single Doses of Orally Administered Investigational Product to Investigate Safety, Tolerability, and Pharmacokinecs.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 111596
Record Dates: First submitted 2008-10-27; First posted 2008-10-31 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Dyslipidaemias
Keywords: tolerability; pharmacodynamics; pharmacokinetics; safety

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): 6 active 2 placebo
  Interventions: Drug: an undetermined dose of GSK1292263
- Cohort 2 (Experimental): 9 active 3 placebo
  Interventions: Drug: ascending dose of GSK1292263
- Cohort 3 (Experimental): Optional cohort
  Interventions: Drug: ascending dose of GSK1292263
- Cohort 4 (Experimental): 12 active
  Interventions: Drug: ascending dose of GSK1292263
- Cohort 5 (Experimental): 12 active
  Interventions: Drug: ascending dose of GSK1292263

INTERVENTIONS:
Drug: an undetermined dose of GSK1292263 — GSK investigational product or placebo
  Arms: Cohort 1
Drug: ascending dose of GSK1292263 — Ascending dose based on target exposures or placebo
  Arms: Cohort 2
Drug: ascending dose of GSK1292263 — An ascending dose based on target exposure
  Arms: Cohort 3
Drug: ascending dose of GSK1292263 — An ascending dose based on target exposures.
  Arms: Cohort 4
Drug: ascending dose of GSK1292263 — An ascending dose based on target exposure
  Arms: Cohort 5

SUMMARY:
This study is the first study in humans to assess the safety and tolerability of various doses of GSK1292263 alone, and taken with sitigliptan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female between 18 and 55 years of age
* A female subject is eligible to participate if she is of non-childbearing potential
* Male subjects must agree to use one of the contraception methods listed in the protocol
* BMI within the range 20 - 29.9 kg/m2
* Capable of giving written informed consent, which includes compliance with protocol
* QTcB or QTcF < 450msec.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen
* Positive urinary cotinine levels or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of regular alcohol consumption within 6 months of the study
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Unable or unwilling to abstain from caffeine-or xanthine-containing products for 24 hours prior to dosing until the final post-dose assessment at each treatment level.
* Use of illicit drugs.
* Use of alcohol for 24 hours prior to dosing until final post-dose assessment at each treatment level.
* Consumption of red wine, oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final pharmacokinetic and pharmacodynamic blood samples
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing
* Lactating females
* Has a fasting triglyceride level >400mg/dL (4.45mmol/L)
* Has anemia defined by hemoglobin concentration <11.0g/dL for males or <10.0g/dL for females.
* CPK values higher than 2.5 times the upper limit of normal at screening.
* Significant ECG abnormalities
* abnormal vital signs as defined in the
* History of any gastrointestinal or hepatic conditions that could impact absorption of the investigational compound.
* Family history (first or second degree relatives) with a history of hypertrophic cardiomyopathy.
* Family history of torsade de pointes or other ventricular arrhythmias.
* Family history of unexplained sudden death.
* Evidence of early depolarization (e.g., Wolf-Parkinson-White syndrome).
* Has clinically significant rhythm abnormalities identified during 24-hour Screening Holter assessment.
* Subjects who have asthma or a history of asthma
* The subject has participated in a clinical trial and has received an investigational product within a protocol defined period
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 14 days if the drug is a potential enzyme inducer or 5 half-lives prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Subjects who are taking low-dose aspirin for cardiovascular prophylaxis (81mg or less) are eligible to participate in the study, but the aspirin must be discontinued from Screening to the Follow-up visit
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Unwillingness or inability to follow the procedures outlined in the protocol.
* As a result of the medical interview, physical examination, or screening investigations, the investigator considers the subject unfit for the study.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-09-04 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters including adverse events, clinical laboratory, electrocardiogram, and vital signs assessments. | Up to 4 days
Pharmacokinetic parameters, maximum observed plasma drug concentration, time to maximum observe. | Up to 4 days

SECONDARY OUTCOMES:
Pharmacodynamic endpoints | Up to four days.
• Pharmacokinetic parameters following a dose, with and without food, and bioavailability | Up to four days.
Relationships betwen drug exposures and pharmacodynamic parameters, safety, and tolerability, as appropriate. | Up to four days.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111596 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111596?search=study&study_ids=11596#rs
- Available data/document: Statistical Analysis Plan: 111596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register